CLINICAL TRIAL: NCT01022567
Title: Study of Surgical Treatment (Open Appendicectomy) Versus Antibiotic Treatment (Ertapenem) in the Treatment of Acute Uncomplicated Appendicitis
Brief Title: Appendicectomy Versus Antibiotics in the Treatment of Acute Uncomplicated Appendicitis
Acronym: APPAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Oulu University Hospital (Other); Tampere University Hospital (Other); Mikkeli Central Hospital (Other); Jyväskylä Central Hospital (Other); Seinajoki Central Hospital (Other)
Responsible Party: Principal Investigator, Paulina Salminen, MD, PhD, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APPAC
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy; Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Operative treatment (Active Comparator): Regular open appendicectomy
  Interventions: Procedure: Appendicectomy
- Antibiotic treatment (Active Comparator): Ertapenem 1 g i.v. x 1 three days
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Procedure: Appendicectomy — Standard appendicectomy
  Arms: Operative treatment
Drug: Ertapenem — ertapenem 1g x 1 i.v.for three days + after discharge levofloxacin 500 mg 1 x 1 + metronidazole 500 mg 1x3 for 7 days p.o.
  Arms: Antibiotic treatment

SUMMARY:
Appendicectomy has been the treatment of acute appendicitis for over a hundred years. Appendicectomy, however, includes operative and postoperative risks despite being a "routine" operation. At the same time other similar intra-abdominal infections, such as diverticulitis, are treated with antibiotics. There have been some encouraging reports on successful treatment of appendicitis with antibiotics and it has been estimated that operative treatment might be necessary for only 15 - 20 % of patients with acute appendicitis.

The aim of this randomized prospective study is to compare operative treatment (open appendicectomy) with conservative treatment with antibiotics (ertapenem, Invanz). Before randomization acute uncomplicated appendicitis is diagnosed with a CT scan.The hypothesis of the study is that the majority of patients with uncomplicated acute appendicitis can be treated successfully with antibiotics and unnecessary appendicectomies can be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 60 years
* CT scan diagnosed uncomplicated acute appendicitis

Exclusion Criteria:

* Age under 18 years or age over 60 years
* Pregnancy or breast-feeding
* Allergy to contrast media or iodine
* Renal insufficiency
* metformin medication (DM)
* Peritonitis (a perforated appendix)
* Lack of co-operation (unable to give consent)
* A severe other medical condition
* CT-scan: other diagnosis, fecal lithiasis in appendix, perforation, abscess, suspicion of a tumour

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 530 (Actual)
Dates: Start 2009-11; Primary Completion 2012-06 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, MD, PhD, Principal Investigator — Department of surgery, Turku University Hospital
Locations (6):
- Finland (6):
  - Keski-Suomi Central Hosptal, Jyväskylä
  - Mikkeli Central Hospital, Mikkeli
  - Oulu University Hospital, Oulu
  - Seinäjoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paajanen H, Gronroos JM, Rautio T, Nordstrom P, Aarnio M, Rantanen T, Hurme S, Dean K, Jartti A, Mecklin JP, Sand J, Salminen P. A prospective randomized controlled multicenter trial comparing antibiotic therapy with appendectomy in the treatment of uncomplicated acute appendicitis (APPAC trial). BMC Surg. 2013 Feb 8;13:3. doi: 10.1186/1471-2482-13-3. PMID 23394263
- [Result] Salminen P, Paajanen H, Rautio T, Nordstrom P, Aarnio M, Rantanen T, Tuominen R, Hurme S, Virtanen J, Mecklin JP, Sand J, Jartti A, Rinta-Kiikka I, Gronroos JM. Antibiotic Therapy vs Appendectomy for Treatment of Uncomplicated Acute Appendicitis: The APPAC Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2340-8. doi: 10.1001/jama.2015.6154. PMID 26080338
- [Derived] Salminen P, Salminen R, Kallio J, Hurme S, Nordstrom P, Rantanen T, Paajanen H, Aarnio M, Mecklin JP, Sand J, Gronroos JM, Rautio T. Antibiotic Therapy for Uncomplicated Acute Appendicitis: Ten-Year Follow-Up of the APPAC Randomized Clinical Trial. JAMA. 2026 Jan 21. doi: 10.1001/jama.2025.25921. Online ahead of print. PMID 41563747
- [Derived] Selanne L, Hurme S, Sippola S, Rautio T, Nordstrom P, Rantanen T, Pinta T, Ilves I, Mattila A, Savela EL, Rintala J, Paajanen H, Gronroos J, Haijanen J, Salminen P. Prognostic factors associated with primary non-responsiveness to antibiotics and appendicitis recurrence for CT-diagnosed uncomplicated acute appendicitis: secondary analysis of two randomized clinical trials. Br J Surg. 2025 Jul 3;112(7):znaf143. doi: 10.1093/bjs/znaf143. PMID 40741675
- [Derived] Sippola S, Haijanen J, Viinikainen L, Gronroos J, Paajanen H, Rautio T, Nordstrom P, Aarnio M, Rantanen T, Hurme S, Mecklin JP, Sand J, Jartti A, Salminen P. Quality of Life and Patient Satisfaction at 7-Year Follow-up of Antibiotic Therapy vs Appendectomy for Uncomplicated Acute Appendicitis: A Secondary Analysis of a Randomized Clinical Trial. JAMA Surg. 2020 Apr 1;155(4):283-289. doi: 10.1001/jamasurg.2019.6028. PMID 32074268
- [Derived] Salminen P, Tuominen R, Paajanen H, Rautio T, Nordstrom P, Aarnio M, Rantanen T, Hurme S, Mecklin JP, Sand J, Virtanen J, Jartti A, Gronroos JM. Five-Year Follow-up of Antibiotic Therapy for Uncomplicated Acute Appendicitis in the APPAC Randomized Clinical Trial. JAMA. 2018 Sep 25;320(12):1259-1265. doi: 10.1001/jama.2018.13201. PMID 30264120
- [Derived] Niiniviita H, Salminen P, Gronroos JM, Rinta-Kiikka I, Hurme S, Kiljunen T, Kulmala J, Teras M, Sippola S, Virtanen J. LOW-DOSE CT PROTOCOL OPTIMIZATION FOR THE ASSESSMENT OF ACUTE APPENDICITIS: THE OPTICAP PHANTOM STUDY. Radiat Prot Dosimetry. 2018 Jan 1;178(1):20-28. doi: 10.1093/rpd/ncx070. PMID 28591824

RESULTS

PARTICIPANT FLOW:
Groups:
- Appendectomy: Open appendectomy
- Antibiotic Therapy: Ertapenem 1 g x 1 for three days followed by levofloxacin 500 mg x 1 combined with metronidazole 500 mg x 3 for seven days.
Period: Overall Study
Arm/Group | Appendectomy | Antibiotic Therapy
Started | 273 | 257
Completed | 272 | 242
Not Completed | 1 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Operative Treatment | Antibiotic Treatment | Total
Number analyzed (Participants) | 273 | 257 | 530
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 273 | 257 | 530
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | 99 | 102 | 201
  Male | 174 | 155 | 329
Region of Enrollment [Number; unit: participants]
  Finland | 273 | 257 | 530

OUTCOME MEASURES:

1. Primary Outcome: The Success of Antibiotic and Surgical Treatment in the Treatment of Acute Uncomplicated Appendicitis
Description: A successful treatment is determined by resolution of the appendicitis by means of the assigned treatment.
Time Frame: Up to 10 years
Population: Treatment success
Measure: Number (95% Confidence Interval); unit: percentage of successful treatment
Arm/Group | Appendectomy | Antibiotic Therapy
Number analyzed (Participants) | 273 | 257
percentage of successful treatment | 99.6 [98.0 to 100.0] | 72.7 [66.8 to 78.0]

2. Secondary Outcome: The Possible Complications, Morbidity and Mortality of Operative and Conservative Treatment
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: The Direct and Indirect Costs of Both Treatment Arms
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: The Recurrence of Conservatively Treated Appendicitis
Time Frame: up to 10 years
Reporting Status: Not Posted, anticipated posting 2022-06

ADVERSE EVENTS:
Arm/Group | Appendectomy | Antibiotic Therapy
Serious Adverse Events (participants affected / at risk) | 0/273 | 0/257
Other Adverse Events (participants affected / at risk) | 45/273 | 6/257
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Appendectomy (N=273) | Antibiotic Therapy (N=257)
Overall morbidity (Infections and infestations) | 45 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No